CLINICAL TRIAL: NCT05464121
Title: A Blended Intervention for Adjustment Disorder: Feasibility Trial and Preliminary Effectiveness.
Brief Title: A Blended Intervention for Adjustment Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UJaumeI_AjD_Blended
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Adjustment Disorders
Keywords: Adjustment Disorders; Internet-based treatment; Blended intervention; Feasibility; Videoconferencing
MeSH Terms: conditions — Adjustment Disorders | interventions — Troleandomycin

STUDY DESIGN:
Intervention Model Description: Patients will be assessed for eligibility and if they meet the inclusion criteria they will be assigned to the single treatment group (single arm). All patients will receive the same blended intervention that combines the self-applied online TAO program with videoconferencing sessions with a therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blended intervention for AjD. (Experimental): Blended intervention for AjD. Main components: psychoeducation, techniques for regulating emotions, exposure, problem-solving techniques, Mindfulness, acceptance and elaboration of the stressful event, positive psychology strategies and relapse prevention.
  Interventions: Behavioral: • Blended treatment for AjD combining a self-applied Internet-based program (TAO) with face-to-face sessions via videoconference.

INTERVENTIONS:
Behavioral: • Blended treatment for AjD combining a self-applied Internet-based program (TAO) with face-to-face sessions via videoconference. — The self-applied Internet-based program called TAO is accessible online from the platform https://psicologiaytecnologia.labpsitec.es. It is organised into 7 sequential modules of approximately 60 minutes. The patient will do a treatment module every 10-12 days, plus an individual session via videoconference with a therapist (approximately 20-30 minutes long). During these sessions, the therapist will explain the main contents of each module, resolve doubts and motivate the patient to continue with the therapy. It takes about 12 weeks to complete the intervention.
  TAO is the optimised version of the original intervention protocol for AjD developed by Botella et al. by Botella et al. (2008) and includes the following therapeutic components: psychoeducation, emotion regulation techniques, exposure, problem-solving techniques, Mindfulness, acceptance and elaboration of the stressful event, positive psychology strategies and relapse prevention.

SUMMARY:
The aim of this study is to evaluate the feasibility (including usability and satisfaction) and preliminary effectiveness of a blended intervention for Adjustment Disorder. This intervention combines a self-applied Internet-based program (TAO) with face-to-face sessions with a therapist via videoconference.

DETAILED DESCRIPTION:
Adjustment disorder (AjD) is one of the most commonly diagnosed disorders in clinical practice. However, although there is still no evidence-based treatment for this problem, Cognitive Behavioral Therapy (CBT) is the most studied. Internet-based treatments emerge as an alternative to reach more people in need while reducing intervention costs. However, high drop-out rates in this format highlight the need to develop new ways of delivering treatments. The present study aims to test a blended treatment for AjD that combines a self-applied CBT programme online (TAO: Adjustment Disorder Online) with face-to-face sessions with a therapist via videoconference every 10-12 days. Only one treatment group has been included and patients will be evaluated at pre-treatment, post-treatment and follow-up (3 and 12 months).

The study will be conducted following the extension of the Consolidated Standards of Reporting Trials (CONSORT) statement for pilot and feasibility studies (Eldridge et al., 2016), the Consolidated Standards of Reporting Trials of Electronic and Mobile Health Applications and online TeleHealth guidelines (Eysenbach, 2011), and the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines (Chan et al., 2013a; 2013b).

Specific objectives of the study include: (1) To analyse the feasibility of different recruitment and data collection methods (e.g., how broad or restrictive are the eligibility criteria, how willing are patients to participate, time needed to collect data), (2) To explore reasons for non-participation and drop-outs from treatment, (3) To assess patient satisfaction and acceptance of treatment (both quantitatively and qualitatively), (4) In addition, as a secondary objective to explore the potential effectiveness of the treatment at post-treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Meeting diagnostic criteria for Adjustment Disorder based on the International Classification of Diseases 11 edition (ICD-11).
* Exceed the cut-off point of 47.5 on the Adjustment Disorder New Module-20 scale (ADNM-20; Lorenz et al., 2016).
* Sign an informed consent.
* Ability to understand and read Spanish.
* Ability to use a computer and having access to the Internet.
* Having an e-mail address.

Exclusion Criteria:

* Presence of risk of suicide or self-destructive behaviors.
* Presence of another severe mental disorder (substance abuse or dependence, psychotic disorder, dementia, bipolar disorder or personality disorder).
* Receiving other psychological treatment during the study for AjD.
* An increase and/or change in the medication during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Participants' adherence to the intervention. | At post-treatment (approximately 12 weeks from the beginning).
  Drop-outs rates (and reasons), number of modules completed, number of times participants enter treatment, time spent in treatment and whether they do reviews.
Expectations and Satisfaction Questionnaire adapted from Borkovec and Nau (1972). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  This questionnaire consists of two different scales. Both include 6 items with a response scale ranging from 0 (not at all) to 10 (completely). One of the scales refers to the expectations about the treatment and it is administered before starting the treatment once an explanation about it has been carried out. The other scale refers to the patients' opinion once they have finished the intervention.
Opinion Questionnaire about the intervention | At post-treatment (approximately 12 weeks from the beginning).
  It assesses participants' opinion about TAO online program, the videoconference sessions with the therapist and the blended format. The questions refer to the satisfaction and usefulness of these components using a response scale from 0 to 10 and open-ended opinion questions.
Working Alliance Inventory for guided Internet Interventions (WAI-I) adapted from Horvath and Greenberg (1989). | At post-treatment (approximately 12 weeks from the beginning).
  The WAI-I scale assesses the different components of therapeutic alliance according to Bordin (1979). This version is adapted for internet-based treatments and consists of 12 items with a response scale from 1 (never) to 7 (always).
Usability System Scale (SUS; Bangor et al., 2008; Brooke,1996). | At post-treatment (approximately 12 weeks from the beginning).
  This scale assesses the usability of a service or product and the acceptance by the users. It consists of 10 items with a response scale ranging from 1 (strongly disagree) to 5 (strongly agree).

SECONDARY OUTCOMES:
Change in Adjustment Disorder New Module-20 (ADNM-20; Einsle et al., 2010). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  Self-report based on ICD-11 diagnostic criteria for AjD. It includes a list of stressful events and another of symptoms. Patients' symptomatology is evaluated in reference to the stressful event that they consider most interferes with them. It uses a response scale from 1 (never) to 4 (frequently). Higher scores indicate greater symptomatology. Lorenz et al. (2016) suggest that a cut off at 47.5 can differentiate between people with low and high risk of AjD.
Change in the Loss and Stress Inventory (IEP) (Quero et al., 2019). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  The IEP consists of 17 items that assess the intensity with which a situation or person lost as a result of the stressful event interferes with the patient's life. It uses a response scale from 0 (never) to 4 (always).
Change in the Positive and Negative Affect Scale (PANAS trait) (Watson et al., 1988; Díaz-García et al., 2020). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  The PANAS assesses two dimensions of mood (positive affect and negative affect). It consists of 20 items describing different emotions or feelings. The patient must respond to the extent to which he or she usually feels the way each expression, using a response scale from 1 (not at all or hardly at all) to 5 (very much).
Change in the Posttraumatic Growth Inventory (PTGI) (Tadeschi and Calhoun,1996; Weiss et al., 2006). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  This measure includes 21 items that assess positive psychological change following an adverse or traumatic experience. It uses a response scale ranging from 0 (I did not experience this change as a result of the crisis) to 5 (I experienced this change to a great extent).
Change in the Overall Anxiety Severity and Impairment Scale (OASIS) (Norman et al., 2006; González-Robles et al., 2018). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  The OASIS measures the frequency and severity of anxiety symptoms, as well as the degree of avoidance and interference. It consists of 5 items with a response scale from 0 to 4. Higher scores indicate greater severity or frequency of symptomatology.
Change in the Overall Depression Severity and Impairment Scale (ODSIS; Norman et al., 2006; Mira et al., 2019). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  The ODSIS measures the frequency and severity of depressive symptoms, as well as the degree of avoidance and interference. It consists of 5 items with a response scale from 0 to 4. One additional item has been included to assess suicide ideation. Higher scores indicate greater severity or frequency of symptomatology.

OTHER OUTCOMES:
Change in efficacy measures after each treatment module. | After each treatment module (i.e. 7 times) for approximately 12 weeks.
  First, patients answer questions about their mood. They are asked to select the face with the emotional expression that best reflects how they are feeling at that moment. Then, they are presented with a list of emotions and must indicate the extent to which they feel each emotion using a scale ranging from "not at all" to "totally". Finally, they are asked how they feel at the end of the module compared to how they felt before they started it. After these questions, changes in self-efficacy, acceptance of the stressful event, openness to future experiences and satisfaction with the module are assessed using a response scale from 0 to 10.
Change in the Purpose-in-Life Test-10 Items (PIL-10) (Crumbaugh and Maholick, 1964; García-Alandete et al., 2013). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  This 10-item instrument assesses different aspects of meaning in life. It uses a response scale from 1 to 7, with higher scores indicating greater meaning of life.
Change in the Quality of Life Inventory (QLI) (Mezzich et al., 1986; Mezzich et al., 2000). | At pre-treatment (before starting the intervention), at post-treatment (approximately 12 weeks from the beginning), and follow-ups (3 and 12 months).
  This measure includes 10 items that assess patients' quality of life in different areas and globally. It uses a response scale from 1 (poor) to 10 (excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, Ph.D, Principal Investigator — Department of Basic, Clinical Psychology and Psychobiology, Universitat Jaume I, Castellón, Spain; Pim Cuijpers, Ph.D, Study Director — Amsterdam Public Health Research Institute, Amsterdam, The Netherlands; Sara Fernández Buendía, Ph.D student, Study Chair — Department of Basic, Clinical Psychology and Psychobiology, Universitat Jaume I, Castellón, Spain
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bachem R, Maercker A. Self-help interventions for adjustment disorder problems: a randomized waiting-list controlled study in a sample of burglary victims. Cogn Behav Ther. 2016 Sep;45(5):397-413. doi: 10.1080/16506073.2016.1191083. Epub 2016 Jun 14. PMID 27299909
- [Background] Botella, C., Baños, R. M., & Guillén, V. (2008). Una propuesta de tratamiento para los Trastornos Adaptativos: Creciendo en la adversidad. In C. Vázquez, & G. Hervás (Eds.), Psicología Positiva Aplicada. Bilbao: DDB.
- [Background] Cucciare, M. A., Weingardt, K. R., & Villafranca, S. (2008). Using blended learning to implement evidence-based psychotherapies. Clinical Psychology: Science and Practice, 15(4), 299-307. https://doi.org/10.1111/j.1468-2850.2008.00141.x
- [Background] Eimontas J, Rimsaite Z, Gegieckaite G, Zelviene P, Kazlauskas E. Internet-Based Self-Help Intervention for ICD-11 Adjustment Disorder: Preliminary Findings. Psychiatr Q. 2018 Jun;89(2):451-460. doi: 10.1007/s11126-017-9547-2. PMID 29124500
- [Background] Leterme AC, Behal H, Demarty AL, Barasino O, Rougegrez L, Labreuche J, Duhamel A, Vaiva G, Servant D. A blended cognitive behavioral intervention for patients with adjustment disorder with anxiety: A randomized controlled trial. Internet Interv. 2020 May 25;21:100329. doi: 10.1016/j.invent.2020.100329. eCollection 2020 Sep. PMID 32523873
- [Background] Lindsater E, Axelsson E, Salomonsson S, Santoft F, Ejeby K, Ljotsson B, Akerstedt T, Lekander M, Hedman-Lagerlof E. Internet-Based Cognitive Behavioral Therapy for Chronic Stress: A Randomized Controlled Trial. Psychother Psychosom. 2018;87(5):296-305. doi: 10.1159/000490742. Epub 2018 Jul 24. PMID 30041167
- [Background] Moser C, Bachem R, Berger T, Maercker A. ZIEL: Internet-Based Self-Help for Adjustment Problems: Results of a Randomized Controlled Trial. J Clin Med. 2019 Oct 11;8(10):1655. doi: 10.3390/jcm8101655. PMID 31614528
- [Background] Quero S, Moles M, Campos D, Andreu-Mateu S, Banos RM, Botella C. An adaptive virtual reality system for the treatment of adjustment disorder and complicated grief: 1-year follow-up efficacy data. Clin Psychol Psychother. 2019 Mar;26(2):204-217. doi: 10.1002/cpp.2342. Epub 2018 Nov 22. PMID 30328216
- [Background] Rachyla I, Mor S, Cuijpers P, Botella C, Castilla D, Quero S. A guided Internet-delivered intervention for adjustment disorders: A randomized controlled trial. Clin Psychol Psychother. 2021 Mar;28(2):313-324. doi: 10.1002/cpp.2518. Epub 2020 Oct 2. PMID 32959481
- [Background] Schuster R, Fichtenbauer I, Sparr VM, Berger T, Laireiter AR. Feasibility of a blended group treatment (bGT) for major depression: uncontrolled interventional study in a university setting. BMJ Open. 2018 Mar 12;8(3):e018412. doi: 10.1136/bmjopen-2017-018412. PMID 29530905
- [Derived] Fernandez-Buendia S, Cuijpers P, Grimaldos J, Diaz-Garcia A, Palau-Batet M, Quero S. A blended intervention for adjustment disorder: Study protocol for a feasibility trial. Internet Interv. 2024 Jan 22;35:100715. doi: 10.1016/j.invent.2024.100715. eCollection 2024 Mar. PMID 38313142